CLINICAL TRIAL: NCT04198194
Title: Apple Heart & Movement Study
Status: Active, not recruiting | Type: Observational
Sponsor: Apple Inc. (Industry)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Calum A. MacRae, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2019P002257
Record Dates: First submitted 2019-11-13; First posted 2019-12-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Prevention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with events: Individuals who have experienced any of the listed outcomes
  Interventions: Diagnostic Test: Predictors of events
- Participants without events: Individuals who have not experienced any of the listed outcomes

INTERVENTIONS:
Diagnostic Test: Predictors of events — Apple Heart & Movement Study in Apple Research app
  Groups: Participants with events

SUMMARY:
This study will look for factors that affect heart health and potentially cause deterioration in mobility or heart function. Participant's Apple Watch and iPhone can help researchers gain a better understanding of potential early warning signs. This can lead to new interventions and products that will help millions lead longer, healthier, and more active lives.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old (at least 19 years old in Alabama and Nebraska, at least 21 years old in Puerto Rico);
* Live in the United States of America;
* Have an iPhone;
* Have an Apple Watch (Series 1 or later) at the time of enrollment;
* Have the Apple Research app installed on your iPhone;
* Be comfortable communicating in written and spoken English;
* Not share your iCloud account, iPhone, or Apple Watch with anyone else;
* Be willing and able to provide informed consent to participate in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will self-enroll in this trial, if they meet inclusion criteria, and there will be no active recruitment of any particular population. Invitation to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Chronic Disease Events | quarterly (every 90 days) through study completion (up to 5 years)
  Change in number of participants with incident cardiovascular disease events (including myocardial infarction, coronary revascularization, heart failure hospitalization, stroke/TIA hospitalization, atrial fibrillation, and atrial fibrillation hospitalization), fall events, and other hospitalizations, assessed by patient report.

CONTACTS AND LOCATIONS:
Overall Officials: Calum A MacRae, MD, PhD, Principal Investigator — cmacrae@bwh.harvard.edu; Angela M Spillane, Study Director — amspillane@bwh.harvard.edu
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No